CLINICAL TRIAL: NCT00164255
Title: Efficacy of Intermittent Sulfadoxine-Pyrimethamine and Sulfadoxine-Pyrimethamine + Artesunate Treatment in the Prevention of Malaria in Pregnancy in an Area With Chloroquine-Resistant Plasmodium Falciparum
Brief Title: Efficacy of Combination Therapy for Prevention of Effects of Malaria During Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ifakara Health Research and Development Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCID-3807; UR3/CCU018969-01
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Malaria
Keywords: malaria; birthweight; placental malaria; intermittent protective treatment; sulfadoxine/ pyrimethamine; artesuate; combination therapy; Pregnancy
MeSH Terms: conditions — Malaria; Birth Weight | interventions — fanasil, pyrimethamine drug combination; Sulfadoxine; Pyrimethamine; Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sulfadoxine/pyrimethamine
Drug: sulfadoxine/pyrimethamine plus artesunate

SUMMARY:
This study is an investigation to compare the efficacy of two different intermittent sulfadoxine/pyrimethamine (SP) treatment regimens and intermittent sulfadoxine/pyrimethamine (SP) + artesunate (SP/AS) treatment of HIV negative and positive mothers in clearing placental parasitemia at delivery. If intermittent protective SP/AS treatment is equally efficacious and safe as intermittent protective SP, such a regimen could be adapted for programmatic use as a potentially more durable alternative to SP monotherapy in areas of increasing SP resistance.

ELIGIBILITY:
Inclusion Criteria:

* Women 15 years of age or older
* First or second pregnancy between 16 and 36 weeks gestation

Exclusion Criteria:

* Pregnancy prior to 16 weeks or after 36 weeks gestation
* Third or later pregnancy;
* Report previous allergic reactions to SP, AS, or unknown antimalarials;
* If the distance to their home is too great or too inaccessible for follow-up;
* Child's father refuses the woman's participation

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1614 (Actual)
Dates: Start 2003-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
placental parasitemia
reported or noted adverse reactions

SECONDARY OUTCOMES:
parasitemia at delivery (maternal peripheral, placental and cord)
maternal illness
birth weight
gestational age
fetal and infant health
impact of maternal HIV infection on efficacy of malaria prevention during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: John MacArthur, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention; Salim Abdulla, MD, PhD, Principal Investigator — Ifakara Health Research and Development Centre
Locations (2):
- Tanzania (2):
  - Kibaoni Health Centre, Ifakara, Kilombero District
  - St Francis Designated District Hospital, Ifakara, Kilombero District

REFERENCES:
- [Derived] Pons-Duran C, Wassenaar MJ, Yovo KE, Marin-Carballo C, Briand V, Gonzalez R. Intermittent preventive treatment regimens for malaria in HIV-positive pregnant women. Cochrane Database Syst Rev. 2024 Sep 26;9(9):CD006689. doi: 10.1002/14651858.CD006689.pub3. PMID 39324693